CLINICAL TRIAL: NCT03659461
Title: Comparative Study of Incretin System in Three Ethnic Groups With Abnormal Glucose Tolerance
Brief Title: Glucagon-like Peptide-1 Levels, Insulin Resistance and Insulin Sensitivity Index in Type 2 Diabetes Mellitus
Acronym: GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Chong Shiau Chin, Pharmacist, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKM-22
Record Dates: First submitted 2018-08-29; First posted 2018-09-06 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low GLP-1 arm (Experimental): Subjects are required to take oral 100mg Sitagliptin (Januvia) daily before breakfast for 12 weeks. 100mg is the recommended treatment dose. During the treatment with Januvia, subjects are not allowed to take any other medications except metformin
  Interventions: Drug: Sitagliptin
- normal GLP-1 arm (Active Comparator): Subjects are required to take oral 100mg Sitagliptin ( Januvia) daily before breakfast for 12 weeks. 100mg is the recommended treatment dose. During the treatment with Januvia, subjects are not allowed to take any other medications except metformin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — oral 100mg Sitagliptin daily will be given for 12 weeks. Subjects are required to undergo OGTT pre and post treatment.

SUMMARY:
This study is conducted to examine GLP-1, insulin resistance and insulin sensitivity portfolio in Malay, Chinese and Indian populations in Malaysia and to study the effect of DPPIV inhibitor in T2DM patients with different GLP-levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are newly diagnosed of T2DM according to World Health Organisation criteria) and do not receive any glucose-lowering drugs
* Subjects with normal glucose tolerance test according to World Health Organisation criteria which is carried out immediately before inclusion in the study
* Subjects who are willing to participate and sign the informed consent form

Exclusion Criteria:

* Patients with pre-existing T2DM
* Patients with family history of diabetes
* Patients receiving glucose-lowering medications
* Patients with anemia, abnormal serum creatinine level, macroalbuminuria, proliferative retinopathy, impaired liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
change in blood glucose load response to sitagliptin | pre-treatment of sitagliptin and post 12-week treatment of sitagliptin
  change from blood glucose response at 12 weeks
change in blood insulin response to sitagliptin | pre-treatment of sitagliptin and post 12-week treatment of sitagliptin
  change from blood insulin response at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kamaruddin Nor Azmi, Study Director — National University of Malaysia; Shiau Chin Chong, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Sultan Ismail, Johor Bahru, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided